CLINICAL TRIAL: NCT05710055
Title: A Randomized, Double-blind, Controlled Trial to Evaluate the Efficacy on Overweight With Oral Supplemenation of Probiotics and Prebiotics
Brief Title: The Efficacy on Overweight With Oral Supplemenation of Probiotics and Prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Precision Health Food Technology Co. Ltd., (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-SM-12-WL-001
Record Dates: First submitted 2023-01-05; First posted 2023-02-02 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Overweight
Keywords: Probiotics; Prebiotics; Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study product A (Wonderlab wonder4shape) (Active Comparator): 2g/bottle, containing the following probiotics total dosage 2.0*10^10 CFU:
  * CECT7527, CECT7528, CECT7529, B420, HN019
  * FOS
  * Polydextrose
  * IMO
  Interventions: Dietary Supplement: Study product A (Wonderlab wonder4shape)
- Study product B (Wonderlab wonder4shape) (Active Comparator): 2g/bottle, containing the following probiotics total dosage 2.0*10^10 CFU:
  * B420, HN019, NCFM
  * FOS
  * Polydextrose
  * IMO
  Interventions: Dietary Supplement: Study product B (Wonderlab wonder4shape)
- Study product C (Wonderlab wonder4shape) (Active Comparator): 2g/bottle, containing the following probiotics total dosage 2.0*10^10 CFU:
  * CECT7527, CECT7528, CECT7529, B420, HN019
  * XOS
  * Polydextrose
  * IMO
  Interventions: Dietary Supplement: Study product C (Wonderlab wonder4shape)
- Study product D (Placebo Comparator): 2g/bottle:
  * MD
  * Cucumber powder
  Interventions: Dietary Supplement: Study product D

INTERVENTIONS:
Dietary Supplement: Study product A (Wonderlab wonder4shape) — Partipants in this arm need to consume one bottle (2g) of this product once a day for 3 months
  Arms: Study product A (Wonderlab wonder4shape)
Dietary Supplement: Study product B (Wonderlab wonder4shape) — Partipants in this arm need to consume one bottle (2g) of this product once a day for 3 months
  Arms: Study product B (Wonderlab wonder4shape)
Dietary Supplement: Study product C (Wonderlab wonder4shape) — Partipants in this arm need to consume one bottle (2g) of this product once a day for 3 months
  Arms: Study product C (Wonderlab wonder4shape)
Dietary Supplement: Study product D — Partipants in this arm need to consume one bottle (2g) of this product once a day for 3 months
  Arms: Study product D

SUMMARY:
The goal of this interventional study is to evaluate the efficacy of probiotics with prebiotics on overweight.

200 eligible participants with overweight will be enrolled and randomized to consume four study products for 3 months.

Reseachers will compare the four groups to evaluate whether there is significant improvement on overweight for participants in the study product of probiotics with prebiotics.

DETAILED DESCRIPTION:
This study is a multi-center, four arms, randomized, double-blind controlled trial. 200 Eligible participants of 25 to 45 years old with overweight will be randomized in four equal size groups to receive one of the four products of probiotics with and without prebiotics and consume one bottle once in a day for 3 months. All participants will visit the study site for 3 times, once a month, all relevant clinical data will be captured, and recorded in to CTMS (Clinical Trial Management System). Data will be analyzed and reported after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chinese males or females, age between 25-45;
* Overweight population: BMI 24-27.9;
* Blood lipids in high potential risks but without medication; TG > 5mol/L, LDL >= 3.4 mmol/L, TC >= 5.2 mmol/L.
* Understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate;
* Agree to avoid medication treatment for weight management, including blood lipids and sugar control.

Exclusion Criteria:

* Have used any medication for weight management at least one month before this study.
* Subject having done plastic surgery for weight management.
* Be involved in any aspect of test administration, i.e., evaluating or overseeing activities related to product.
* Have participated in any clinical study involving the test sites within the previous 6 months, or is subject participating in any clinical study concurrently.
* Have a history of any type of metabolic syndrome, including but not limited to any type of diabetes, obesity and heart disease.
* Have a history of any disease or the presence of health condition on the study sites that the Investigator feels would interfere with the study.
* Be taking antihistamines (> 3x/week) or anti-inflammatory (> 8x/week) on a regular basis, or has the subject taken systemic or topical steroidal medications within 4 weeks of study enrollment.
* Have any of the following conditions or factors that the investigator believes may affect the response of the skin or the interpretation of the test results, including, but not limited to, pregnancy, lactation and hepatitis.
* Have any cuts/abrasions on the test site at baseline.
* The subject is an employee of sponsor or the site conducting the study.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change of Weight | baseline day 0, day 60
  Change of Weight in Kg by Inbody S10 from baseline to 2 months

SECONDARY OUTCOMES:
Blood lipids - Total Cholesterol Level | baseline day 0, visit 1 day 30, visit 2 day 60, visit 3 day 90
  Blood lipids - Total Cholesterol level of blood test in mmol/L and range of 0.56-17mmol/L for each visit interval
Blood Sugar Level | baseline day 0, visit 1 day 30, visit 2 day 60, visit 3 day 90
  Blood sugar level of blood test in mmol/L and range of 3.9-6.1mmol/L for each visit interval
Blood Hormone - Leptin Level | baseline day 0, visit 1 day 30, visit 2 day 60, visit 3 day 90
  Blood hormone - Leptin level of blood test in ng/mL and range 0.5-15.2ng/mL for each visit interval
Blood Hormone - Adiponectin Level | baseline day 0, visit 1 day 30, visit 2 day 60, visit 3 day 90
  Blood hormone - Adiponectin level of blood test in ug/mL and range of 2-37ug/mL for each visit interval
Blood inflammation | baseline day 0, visit 1 day 30, visit 2 day 60, visit 3 day 90
  Blood inflammation (Zonulin, ApoB-48, hsCRP, LPS, sCD14, IL-6, MCP-1, Angptl4) for each visit interval
Feces SCFA | baseline day 0, visit 1 day 30, visit 2 day 60, visit 3 day 90
  Feces SCFA for each visit interval
Feces sIgA | baseline day 0, visit 1 day 30, visit 2 day 60, visit 3 day 90
  Feces sIgA for each visit interval
Liver function test | baseline day 0, visit 1 day 30, visit 2 day 60, visit 3 day 90
  Liver function test for each visit interval

CONTACTS AND LOCATIONS:
Overall Officials: Weixing Wang, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Ai'er Hospital, Shanghai, Shanghai Municipality
  - SPRIM Central Lab, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suzumura EA, Bersch-Ferreira AC, Torreglosa CR, da Silva JT, Coqueiro AY, Kuntz MGF, Chrispim PP, Weber B, Cavalcanti AB. Effects of oral supplementation with probiotics or synbiotics in overweight and obese adults: a systematic review and meta-analyses of randomized trials. Nutr Rev. 2019 Jun 1;77(6):430-450. doi: 10.1093/nutrit/nuz001. PMID 30924853
- [Background] Rouxinol-Dias AL, Pinto AR, Janeiro C, Rodrigues D, Moreira M, Dias J, Pereira P. Probiotics for the control of obesity - Its effect on weight change. Porto Biomed J. 2016 Mar-Apr;1(1):12-24. doi: 10.1016/j.pbj.2016.03.005. Epub 2016 Mar 1. PMID 32258541
- [Background] Perna S, Ilyas Z, Giacosa A, Gasparri C, Peroni G, Faliva MA, Rigon C, Naso M, Riva A, Petrangolini G, A Redha A, Rondanelli M. Is Probiotic Supplementation Useful for the Management of Body Weight and Other Anthropometric Measures in Adults Affected by Overweight and Obesity with Metabolic Related Diseases? A Systematic Review and Meta-Analysis. Nutrients. 2021 Feb 19;13(2):666. doi: 10.3390/nu13020666. PMID 33669580
- [Background] Michael DR, Davies TS, Jack AA, Masetti G, Marchesi JR, Wang D, Mullish BH, Plummer SF. Daily supplementation with the Lab4P probiotic consortium induces significant weight loss in overweight adults. Sci Rep. 2021 Jan 6;11(1):5. doi: 10.1038/s41598-020-78285-3. PMID 33408364
- [Background] Nasiri G, Bastani A, Haji-Aghamohammadi AA, Nooshabadi MR, Shahmirzalou P, Haghighian HK. Effects of probiotic and alpha-lipoic acid supplements, separately or in combination on the anthropometric indicators and maintenance of weight in overweight individuals. Clin Nutr ESPEN. 2021 Feb;41:242-248. doi: 10.1016/j.clnesp.2020.12.007. Epub 2020 Dec 30. PMID 33487271
- [Background] Dechelotte P, Breton J, Trotin-Picolo C, Grube B, Erlenbeck C, Bothe G, Fetissov SO, Lambert G. The Probiotic Strain H. alvei HA4597(R) Improves Weight Loss in Overweight Subjects under Moderate Hypocaloric Diet: A Proof-of-Concept, Multicenter Randomized, Double-Blind Placebo-Controlled Study. Nutrients. 2021 Jun 1;13(6):1902. doi: 10.3390/nu13061902. PMID 34205871
- [Background] Stenman LK, Lehtinen MJ, Meland N, Christensen JE, Yeung N, Saarinen MT, Courtney M, Burcelin R, Lahdeaho ML, Linros J, Apter D, Scheinin M, Kloster Smerud H, Rissanen A, Lahtinen S. Probiotic With or Without Fiber Controls Body Fat Mass, Associated With Serum Zonulin, in Overweight and Obese Adults-Randomized Controlled Trial. EBioMedicine. 2016 Nov;13:190-200. doi: 10.1016/j.ebiom.2016.10.036. Epub 2016 Oct 26. PMID 27810310
- [Background] Magro DO, de Oliveira LM, Bernasconi I, Ruela Mde S, Credidio L, Barcelos IK, Leal RF, Ayrizono Mde L, Fagundes JJ, Teixeira Lde B, Ouwehand AC, Coy CS. Effect of yogurt containing polydextrose, Lactobacillus acidophilus NCFM and Bifidobacterium lactis HN019: a randomized, double-blind, controlled study in chronic constipation. Nutr J. 2014 Jul 24;13:75. doi: 10.1186/1475-2891-13-75. PMID 25056655
- [Background] Waller PA, Gopal PK, Leyer GJ, Ouwehand AC, Reifer C, Stewart ME, Miller LE. Dose-response effect of Bifidobacterium lactis HN019 on whole gut transit time and functional gastrointestinal symptoms in adults. Scand J Gastroenterol. 2011 Sep;46(9):1057-64. doi: 10.3109/00365521.2011.584895. Epub 2011 Jun 13. PMID 21663486
- [Background] Fuentes MC, Lajo T, Carrion JM, Cune J. Cholesterol-lowering efficacy of Lactobacillus plantarum CECT 7527, 7528 and 7529 in hypercholesterolaemic adults. Br J Nutr. 2013 May 28;109(10):1866-72. doi: 10.1017/S000711451200373X. Epub 2012 Sep 28. PMID 23017585
- [Background] Guerrero-Bonmatty R, Gil-Fernandez G, Rodriguez-Velasco FJ, Espadaler-Mazo J. A Combination of Lactoplantibacillus plantarum Strains CECT7527, CECT7528, and CECT7529 Plus Monacolin K Reduces Blood Cholesterol: Results from a Randomized, Double-Blind, Placebo-Controlled Study. Nutrients. 2021 Apr 6;13(4):1206. doi: 10.3390/nu13041206. PMID 33917503